CLINICAL TRIAL: NCT03479840
Title: Age-Dependent Impact of the SYNTAX-score on Mortality After Percutaneous Coronary Intervention in an All-Comer Population
Brief Title: Age-Dependent Impact of the SYNTAX-score on Mortality
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julinda Mehilli, Prof. Dr. med., LMU Klinikum
Other Study IDs: GEMucI003-16
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; PCI
Keywords: SYNTAX score, PCI, elderly
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing PCI: all-comer population undergoing PCI
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — treatment of coronary arteries and evaluation of SYNTAX score pre and post (to quantify severity of disease)
  Other Names: percutaneous coronary intervention

SUMMARY:
The SYNTAX-score has been proposed as a tool for risk stratification and guiding revascularization therapy in patients with complex coronary artery disease.

There are limited data on the prognostic value of the SYNTAX-score among elderly patients.

Aim of this study was to investigate whether age modifies the impact of the SYNTAX-score on all-cause mortality at 2 years after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
SYNTAX score has been used as a tool to quantify severity of coronary artery disease. Interventional or operative treatment of patients is associated with improvement in SYTAX score after PCI so called residual SYNTAX score. The higher the SYNTAX score value the higher is the mortality. Whereas this is true for both young and old patients is debatable. Therefore we aim to investigate in this registry age-dependent impact of baseline and residual SYNTAX score on 1- and 2-year mortality after PCI

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing PCI at our center

Exclusion Criteria:

* prior coronary artery bypass grafting
* no PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comer population undergoing PCI
Sampling Method: Non-Probability Sample
Enrollment: 1331 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Medium- to long-term Mortality | 2 years
  Overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — LMU Klinikum
Locations (1):
- Ludwig-Maximilians University, Munich, Germany

IPD SHARING:
Plan to Share IPD: No